CLINICAL TRIAL: NCT01023893
Title: Clinical Diagnostic Evaluation Study of Blood Viscosity, End-Stage Renal Disease, And Mortality
Brief Title: Blood Viscosity, End-Stage Renal Disease, And Mortality (BEAM-1)
Acronym: BEAM-1
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: ProMetrics, Inc. (Industry)
Responsible Party: Daniel Cho, VP Lab Services, ProMetrics
Other Study IDs: PRO-0062-201
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- End-stage renal disease

SUMMARY:
Prospective, real-time observational study of hemodialysis patients treated with erythropoiesis-stimulating agents (ESA) to currently recommended Hgb targets. Subjects will be evaluated dynamically for their blood viscosity status at the beginning and end of the dialysis treatment, and followed prospectively to assess outcomes. Blood specimens will be collected via the subject's hemodialysis port pre- and post-hemodialysis per study assessment visit. Blood will be analyzed at a designated laboratory facility for viscosity over a comprehensive range of shear rates and tested for intradialytic surges in blood viscosity. Subjects will be followed for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* On hemodialysis > 3 months
* On ESA treatment > 3 months
* Mean Hgb 11 g/dL - 12 g/dL (based on at least 3 Hgb results during the previous 8 weeks)
* Latest Hgb 10.5 g/dL - 12.5 g/dL (measured within 1 week of study)

Exclusion Criteria:

* Inability or unwillingness to provide informed consent
* Large variability in interdialytic weight gain (>2 kg difference between low and high weight gain over last month)
* More than 1 missed dialysis treatments in past month
* Recent bleeding
* Blood transfusion within 1 month
* Hematologic disease other than anemia
* Active inflammatory disease
* Active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dialysis clinic
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular mortality | One year

SECONDARY OUTCOMES:
All-cause mortality | One year
Vascular access thrombosis | One year

REFERENCES:
- [Background] Vaisman S, Kensey K, Cho YI. Effect of hemodialysis on whole blood viscosity. Int J Artif Organs. 2009 Jun;32(6):329-35. doi: 10.1177/039139880903200603. PMID 19670184
- [Background] Lowe GD, Lee AJ, Rumley A, Price JF, Fowkes FG. Blood viscosity and risk of cardiovascular events: the Edinburgh Artery Study. Br J Haematol. 1997 Jan;96(1):168-73. doi: 10.1046/j.1365-2141.1997.8532481.x. PMID 9012704